CLINICAL TRIAL: NCT04831008
Title: Comparison of Figure-Of-Eight Suture and Perclose ProGlide Suture-Mediated Closure System in Achieving Hemostasis After a Large Bore Venous Access.
Brief Title: Comparison of Figure-Of-Eight Suture Perclose ProGlide Suture-Mediated Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delray Medical Center (Other)
Collaborators: Florida Atlantic University (Other)
Responsible Party: Principal Investigator, Houman Khalili MD, Principal Investigator, Delray Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-149
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Venous Puncture
Keywords: Perclose Device; Figure-of-eight suture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Figure-of-eight (Active Comparator): Using the figure-of-eight closure technique when closing access for structural heart therapies.
  Interventions: Other: Figure-of-eight suture
- Perclose Device (Active Comparator): Using the Perclose device when closing access for structural heart therapies.
  Interventions: Other: Perclose Device

INTERVENTIONS:
Other: Figure-of-eight suture — Using the figure-of-eight closure technique when closing access for structural heart therapies.
  Arms: Figure-of-eight
Other: Perclose Device — Using the Perclose device when closing access for structural heart therapies.
  Arms: Perclose Device

SUMMARY:
The study proposes to compare specialized closure devices to achieve hemostasis with the Figure-of-eight suture technique.

DETAILED DESCRIPTION:
Procedures where patients requiring large bore venous access will be randomized 1:1 to either the Figure-of-eight suture technique or the Perclose Device to achieve hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* All patients who successfully undergo venous large bore access sheath placement for structural heart procedures.

Exclusion Criteria:

* Patients who do not consent
* Minors or those unable to consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Hemostasis Time | Immediate
  To assess if an additional device use to achieve hemostasis can be avoided after a large bore venous access
Procedure Time | Immediate
Access Site Complication | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Houman Khalili, MD, Principal Investigator — Delray Medical Center; Brijeshwar Maini, Principal Investigator — Delray Medical Center
Locations (1):
- Delray Medical Center, Delray Beach, Florida, United States